CLINICAL TRIAL: NCT01096238
Title: Follow-up of Immunogenicity of Influenza Virus Vaccine, AdimFlu-S (A/H1N1), in Healthy Volunteers After 6 Months
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Huang, Kuo Chin, National Taiwan University Hospital
Other Study IDs: 201002050R
Record Dates: First submitted 2010-03-29; First posted 2010-03-31 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Influenza
Keywords: The immunogenicity of Influenza Virus Vaccine, AdimFlu-S (A/H1N1), in adults after half a year will be analyzed and discussed.
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
In the spring of 2009, a recently emerged novel influenza A (H1N1) virus was first identified in Mexico and USA and it has continued to spread globally. The rapid global spread of a novel influenza A (H1N1) 2009 virus prompted the World Health Organization (WHO), on 11 June 2009, to declare the first influenza pandemic in 41 years. In Taiwan, a clinical study to assess the immunogenicity and safety of Influenza Virus Vaccine, AdimFlu-S (A/H1N1), in healthy volunteers has already been completed. In the previous study, we found that a single 15 mcg HA dose of the AdimFlu-S (A/H1N1) vaccine induces a protective immune response in most adults, including those > 60 years of age (>70%). Our current study aims to follow-up subjects who received Influenza Virus Vaccine, AdimFlu-S (A/H1N1), six months ago. These subjects' serum samples were tested for anti-hemagglutinin (HA) antibodies by hemagglutination inhibition (HAI). The seroconversion is defined as the post-vaccination serum HAI titer had at least 1:40 for subjects who had seronegative pre-vaccination or a four-fold or greater increase in HAI titers for subjects who had seropositive pre-vaccination serum. The immunogenicity of Influenza Virus Vaccine, AdimFlu-S (A/H1N1), in adults after half a year will be analyzed and discussed among the subjects with serum HAI titer had at least 1:40 at least 3 weeks after AdimFlu-S (A/H1N1) injection.

ELIGIBILITY:
Inclusion Criteria:

* subjects with serum HAI titer had at least 1:40 at least 3 weeks after AdimFlu-S (A/H1N1) injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: age>=18 who had AdimFlu-S(A/H1N1) injection
Sampling Method: Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2010-03

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chin Huang, Post Doctor, Principal Investigator — National Taiwan University Hospital